CLINICAL TRIAL: NCT03447223
Title: Gut Microbiome and Serum Metabolome Alterations in Attention-deficit/Hyperactivity Disorder Patients
Brief Title: Gut Microbiome and Serum Metabolome Alterations in ADHD Patients
Acronym: ADHD
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20182002-1
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Attention-deficit/Hyperactivity Disorder
Keywords: Attention-deficit/hyperactivity disorder; circulating metabolites; metagenome
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood samples: serum metabolomics analyses; faeces: gut metagenome analyses
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ADHD-patients: The children and adolescent 6-15 years old with ADHD. Diagnoses of the children with ADHD were made in Xijing Hospital according to criteria described in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV). Children with ADHD had an IQ score above 70.
- Controls-healthy children: Age- and gender- matched healthy 6-15 years old children and adolescent.

SUMMARY:
Host-microbe interactions play a key role in brain development and function and in the etiology of neurodevelopmental disorders. Attention-deficit/hyperactivity disorder (ADHD) is a heterogeneous disorder that affects 1 in 20 children and results in poor life-time outcomes. However, the etiology of ADHD is unclear and its diagnosis and treatment are still challenging. Different factors reported to be associated with the risk of developing ADHD and/or linked to different ADHD manifestations have also been linked to shifts in gut microbiota composition, suggesting a link between the microbiota and the disorder. Here, we will perform a metagenome-wide association study and serum metabolomics profiling in a cohort of control and ADHD, 6-15 years, Chinese individuals. We aim to identify ADHD-associated gut microbial species linked to changes in circulating metabolites. We also aim to find the possible intervention strategy in ADHD by targeting the gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

Diagnoses of the children with ADHD were made in Xijing Hospital according to criteria described in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV). Children with ADHD had an IQ score above 70.

Exclusion Criteria:

Children who had a past history of or were currently affected by neurological diseases, including convulsive disorders or brain damage; or who had any evidence of comorbid psychiatric conditions, such as Tourette's syndrome, IQ below 70, pervasive developmental disorder (autism), bipolar disorder, psychosis, language difficulties or learning disorders (reading disorders, mathematics disorders and disorders of written expression).

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All subjects were drug-naive at the time of recruitment, and the ADHD tests were administered before the subjects were given any medication. The subjects will be recruited from Xijing Hospital and elementary and secondary schools in China.
Sampling Method: Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-05-27 (Actual)

PRIMARY OUTCOMES:
ADHD-associated gut microbial species alterations | 2018-2020
  Gut metagenome analysis with fecal samples

SECONDARY OUTCOMES:
ADHD-associated circulating metabolites alterations | 2018-2020
  Circulation metabonomics analysis with serum samples

CONTACTS AND LOCATIONS:
Overall Officials: Lize Xiong, M.D./Ph.D., Principal Investigator — Professor and President, Xijing Hospital
Locations (1):
- Department of Pediatrics, Xijing Hospital, the Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Result] Sharma A, Couture J. A review of the pathophysiology, etiology, and treatment of attention-deficit hyperactivity disorder (ADHD). Ann Pharmacother. 2014 Feb;48(2):209-25. doi: 10.1177/1060028013510699. Epub 2013 Nov 1. PMID 24259638
- [Result] Aarts E, Ederveen THA, Naaijen J, Zwiers MP, Boekhorst J, Timmerman HM, Smeekens SP, Netea MG, Buitelaar JK, Franke B, van Hijum SAFT, Arias Vasquez A. Gut microbiome in ADHD and its relation to neural reward anticipation. PLoS One. 2017 Sep 1;12(9):e0183509. doi: 10.1371/journal.pone.0183509. eCollection 2017. PMID 28863139
- [Result] Evangelisti M, De Rossi P, Rabasco J, Donfrancesco R, Lionetto L, Capi M, Sani G, Simmaco M, Nicoletti F, Villa MP. Changes in serum levels of kynurenine metabolites in paediatric patients affected by ADHD. Eur Child Adolesc Psychiatry. 2017 Dec;26(12):1433-1441. doi: 10.1007/s00787-017-1002-2. Epub 2017 May 19. PMID 28527020
- See also: Wikipedia — https://en.wikipedia.org/wiki/Attention_deficit_hyperactivity_disorder